CLINICAL TRIAL: NCT00577993
Title: Fludarabine, Mitoxantrone, and Dexamethasone (FND) Plus Chimeric Anti-CD20 Monoclonal Antibody (Rituximab) for Stage IV Indolent Lymphoma
Brief Title: Fludarabine, Mitoxantrone, and Dexamethasone (FND) Plus Rituximab for Lymphoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM97-261; NCI-2010-01566 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Lymphoma
Keywords: Lymphoma; Follicular Lymphoma; Indolent Lymphoma; Fludarabine; Novantrone; Mitoxantrone; Decadron; Dexamethasone; Rituximab; Anti-CD20; IDEC-C2B8; Chimeric Anti-CD20 Antibody; Interferon; Interferon Alpha-2b; IFN; Doxorubicin; Vincristine; Bleomycin; Cyclophosphamide; Etoposide; Cisplatin; Ara-C; Methyl-Prednisolone; Procarbazine; Prednisone; FND
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — fludarabine; Mitoxantrone; Calcium Dobesilate; Dexamethasone; Rituximab; Interferons; Introns; Doxorubicin; Vincristine; Bleomycin; Cyclophosphamide; Etoposide; Cisplatin; Cytarabine; Procarbazine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1: FND + Rituximab Followed by Interferon (Active Comparator): Fludarabine/Novantrone/Decadron + Rituximab Followed by Interferon
  Interventions: Drug: Fludarabine; Drug: Novantrone; Drug: Decadron; Drug: Rituximab; Drug: Interferon
- 2: FND Followed by Interferon & Rituximab (Active Comparator): Fludarabine/Novantrone/Decadron Followed by Interferon & Rituximab
  Interventions: Drug: Fludarabine; Drug: Novantrone; Drug: Decadron; Drug: Rituximab; Drug: Interferon
- 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon (Active Comparator): Cyclophosphamide/Vincristine/Doxorubicin/Bleomycin (1st Sequence) + Rituximab; Etoposide/Cisplatin/Ara-C/Methyl-Prednisol (2nd Sequence); Novantrone/Vincristine/Procarbazine/Prednisone + Rituximab (3rd Sequence) Followed by Interferon
  Interventions: Drug: Novantrone; Drug: Decadron; Drug: Rituximab; Drug: Interferon; Drug: Doxorubicin; Drug: Vincristine; Drug: Bleomycin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Cisplatin; Drug: Ara-C; Drug: Methyl-Prednisolone; Drug: Procarbazine; Drug: Prednisone

INTERVENTIONS:
Drug: Fludarabine — Group 1= 25 mg/m^2 IV over 15 min. Days 2 through 4 for 8 Cycles; Group 2 = 25 mg/m^2 IV over 15 min. Days 1 through 3 for 8 Cycles.
  Other Names: 2-fluoro-Ara Amp
  Arms: 1: FND + Rituximab Followed by Interferon; 2: FND Followed by Interferon & Rituximab
Drug: Novantrone — Group 1 = 10 mg/m^2 IV over 15 min. Day 2 for 8 Cycles; Group 2 = 10 mg/m^2 IV over 15 min. Day 1 for 8 Cycles; Group 3 = 10 mg/m^2 IV over 15 min. Day 2 of 3rd Sequence.
  Other Names: Mitoxantrone
Drug: Decadron — Group 1 = 20 mg IV over 15 min. Days 1 through 5 for 8 Cycles, then Days 1 through 3 Every Month for 1 Year; Group 2 = 20 mg IV over 15 min. Days 1 through 5 for 8 Cycles, then Days 1 through 3 Every Month for 1 Year; Group 3 = 40 mg PO Days 1 through 4 of 1st Sequence; After Completion of 3 Sequences, Days 1 through 3 Every Month for 1 Year.
  Other Names: Dexamethasone
Drug: Rituximab — Group 1 = 375 mg/m^2 IV Days 1 through 8 of Course 1, then Day 1 Only of Cycles 2 through 5; Group 2 = 4 Months after IFN Starts, 375 mg/m^2 IV Once Per Month for 6 Months; Group 3 = 375 mg/m^2 IV Days 1 through 8 of 1st Sequence; 375 mg/m^2 IV Days 1 through 8 of 3rd Sequence.
  Other Names: Chimeric Anti-CD20 Antibody; Anti-CD20; IDEC-C2B8
Drug: Interferon — Group 1 = After Completion of Fludarabine, Novantrone, & Rituximab, IFN 3 mcg/ml/m^2 SQ Days 1 through 14 Each Month for 1 year; Group 2 = After Completion of Fludarabine & Novantrone, IFN 3 mcg/ml/m^2 SQ Days 1 through 14 Each Month for 1 year; Group 3 = After Completion of 3 Sequences, IFN 3 mcg/ml/m^2 SQ Days 1 through 14 Each Month for 1 year.
  Other Names: Interferon Alpha-2b; IFN
Drug: Doxorubicin — 25 mg/m^2 IV Days 2 & 3 of 1st Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Vincristine — .7 mg/m^2 IV Days 2 & 3 of 1st Sequence; 1.4 mg/m^2 IV Day 2 of 3rd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Bleomycin — 5 unit/m^2 IV Days 2 & 3 of 1st Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Cyclophosphamide — 750 mg/m^2 IV Day 2 of 1st Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Etoposide — 40 mg/m^2 IV Days 1 through 4 of 2nd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Cisplatin — 25 mg/m^2 IV Days 1 through 4 of 2nd Sequence
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Ara-C — 1.5 gm/m^2 IV Day 5 of 2nd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Methyl-Prednisolone — 500 mg IV Days 1 through 5 of 2nd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Procarbazine — 100 mg/m^2 PO Days 2 through 11 of 3rd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon
Drug: Prednisone — 100 mg PO Days 1 through 5 of 3rd Sequence.
  Arms: 3: CHOD-Bleo, ESHAP, NOPP + Rituximab Followed by Interferon

SUMMARY:
The goal of this clinical research study is to compare chemotherapy given with rituximab to chemotherapy followed by rituximab. The safety of both treatment schedules will be studied. Laboratory tests of genetic changes in blood and bone marrow before and during the study will also be monitored.

DETAILED DESCRIPTION:
Rituximab is a monoclonal antibody that is designed to attach to leukemia cells and activate a series of events that may cause the cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Mitoxantrone is designed to stop cancer cells from making DNA, which may stop the cells from making more cells.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to MM patients in combination with other chemotherapy to treat cancer.

Study Groups:

If you are found eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. Each group will receive 8 "cycles" of treatment. One (1) cycle will last 28 days.

Group 1:

If you are in Group 1, you will receive the following drugs at the following times. Each study cycle is 28 days:

* Rituximab will be given through a needle in the vein over about 90 minutes on Days 1 and 8 of the first course Cycle 1, and on Day 1 only of Cycles 2-5 of Fludarabine/ Mitoxantrone/ Dexamethasone (FND) treatment.
* Fludarabine will be given through a needle in the vein over about 15 minutes on Days 2-4 of each cycle.
* Mitoxantrone will be given through a needle in the vein over about 15 minutes on Day 2 of each cycle.
* You will take dexamethasone by mouth with water on Days 1-5 of each 28-day cycle (FND).

If you miss any doses of the study drugs, please contact the research staff for instructions.

You will not receive rituximab in Cycles 6-8. When the 8 cycles are finished, you will begin receiving the drug interferon on Days 1-14 each month for 1 year. Dexamethasone will be given on Days 1-3 every month for 1 year.

Patients in group 2 will receive fludarabine on Days 1-3, mitoxantrone on Day 1, and dexamethasone on Days 1-5 of each 28-day cycle. When 8 cycles of treatment are finished, patients will begin receiving the drug interferon on Days 1-14 each month for 1 year. Dexamethasone will be given on Days 1-3 every month for 1 year. About 4 months after interferon treatment starts, patients in group 2 will begin receiving rituximab once a month for 6 months.

Other drugs may be given to help decrease the risk of or ease side effects. Treatment may be delayed or stopped if side effects are severe.

Most of the drugs are given by vein. A catheter (a tube) will be placed in a vein to decrease the number of needle sticks. Dexamethasone may be taken by mouth instead of given by vein.

Some patients in this study, with changes in certain genes will receive different chemotherapy drugs than other patients in the study will. The patients will, like all the other patients, receive rituximab and interferon. But instead of the FND chemotherapy regimen, they will receive a sequence of three regimens, CHOD-Bleo, ESHAP, and NOPP. The drugs in these regimens include: cyclophosphamide, doxorubicin, vincristine, bleomycin, VP-16, Ara-C, cisplatin, mitoxantrone, procarbazine, and corticosteroids (prednisone, methylprednisolone, dexamethasone).

During the study, patients will have blood tests every week. Complete exams will be given in Cycles 2 and 4; patients will return to the clinic for these. Every 2 or 3 cycles, patients will have a chest x-ray and CT scans of the abdomen and pelvis. Bone marrow samples will be taken. Heart function tests (EKG) will be done as needed.

After the study ends, patients will return for checkups every 3 months in the first year, every 4 months in years 2 and 3, and every 6 months in years 4 and 5. After that, checkups will be needed once a year. Blood and bone marrow samples will be taken at these visits.

This is an investigational study. Rituximab is approved by FDA for commercial use. The other drugs used in the study are also approved for commercial use. About 210 patients will take part in the study. All will be enrolled at University of Texas MD Anderson Cancer Center (UTMDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated stage IV indolent B-cell lymphoma [Amendment May 2001: eligibility restricted to follicular lymphoma]
2. Age <76

Exclusion Criteria:

N/A

Max Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 1998-03-16 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 1998 to May 2002
Pre-assignment Details: 35 participants without Bcl Gene rearrangement were not randomized to the study
Groups:
- Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab: Fludarabine,Mitoxantrone, and Dexamethasone (FND) with follow-up Ritux,Flidara,Mitoxan,Dex
- Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND): Fludarabine,Mitoxantrone, and Dexamethasone (FND) with concurrent Ritux,Flidara,Mitoxan,Dex.
- Patients Without Bcl Gene Rearrangement: ATT9 cycles; Rituximab 6 cycles
Period: Overall Study
Arm/Group | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND) | Patients Without Bcl Gene Rearrangement
Started | 85 | 90 | 35
Completed | 78 | 80 | 32
Not Completed | 7 | 10 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Conversion | 2 | 5 | 0
Not completed — Uninsured | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data collected for Patients w/o bcl gene for rearrangement for the Study Specific Measure Indolent Lymphoma Subtype
Groups:
- Patients w/o Bcl Gene Rearrangement: ATT 9 cycles; Rituximab 6 cycles
- Total: Total of all reporting groups
Arm/Group | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND) | Patients w/o Bcl Gene Rearrangement | Total
Number analyzed (Participants) | 78 | 80 | 35 | 193
Age, Continuous [Mean (Full Range); unit: years] | 52 [23 to 76] | 54 [19 to 75] | 51 [33 to 70] | 52 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 34 | 18 | 103
  Male | 27 | 46 | 17 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 13
  Not Hispanic or Latino | 67 | 64 | 27 | 158
  Unknown or Not Reported | 7 | 11 | 4 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 1 | 3 | 11
  White | 63 | 67 | 28 | 158
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 11 | 4 | 22
Region of Enrollment [Number; unit: participants]
  United States | 76 | 77 | 34 | 187
  United Arab Emirates | 0 | 1 | 0 | 1
  China | 0 | 1 | 1 | 2
  Panama | 0 | 1 | 0 | 1
  Malta | 1 | 0 | 0 | 1
  Mexico | 1 | 0 | 0 | 1
Indolent Lymphoma Subtype [Number; unit: participants] — Indolent lymphomas characterized by slow-growing B-cell malignancies: Small lymphocyte (SLL), Malignant Zone (MZL), & Follicular Lymphoma (FL). Population: No data collected for Patients w/o bcl gene for rearrangement for the Study Specific Measure Indolent Lymphoma Subtype
  participants
    FL: number analyzed (Participants) | 78 | 80 | 0 | 158
    FL | 56 | 55 |  | 111
    MZL: number analyzed (Participants) | 78 | 80 | 0 | 158
    MZL | 6 | 12 |  | 18
    SLL: number analyzed (Participants) | 78 | 80 | 0 | 158
    SLL | 16 | 13 |  | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Survival (10 Years) by Treatment
Description: Overall Survival is the time from date of treatment start until date of death due to any cause or last Follow-up within 10 years.
Time Frame: 10 Years
Population: The outcome measures were only being analyzed for the two randomized arms Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab and Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND)
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND)
Number analyzed (Participants) | 78 | 80
Participants | 59 | 58

2. Secondary Outcome: Number of Participants With Progression Free Survival (10 Years) by Treatment
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 10 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND)
Number analyzed (Participants) | 78 | 80
Participants | 59 | 58

ADVERSE EVENTS:
Time Frame: 10 years
Description: Adverse events reported for the 2 randomized arms and not for the participants without bcl gene rearrangement.
Arm/Group | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND)
All-Cause Mortality (participants affected / at risk) | 19/78 | 22/80
Serious Adverse Events (participants affected / at risk) | 67/78 | 77/80
Other Adverse Events (participants affected / at risk) | 67/78 | 77/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab (N=78) | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND) (N=80)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 15 | 12
Fever (General disorders) | 1 | 3
Neutropenic Fever (Blood and lymphatic system disorders) | 2 | 4
Infection (Infections and infestations) | 8 | 15
Nausea/Emesis (Gastrointestinal disorders) | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 67 | 77
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 23
Anemia (Blood and lymphatic system disorders) | 10 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine,Mitoxantrone, and Dexamethasone (FND)-Rituximab (N=78) | Rituximab- Fludarabine,Mitoxantrone, and Dexamethasone (FND) (N=80)
Abdominal Pain (Gastrointestinal disorders) | 21 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 35
Fatigue (General disorders) | 44 | 48
Fever (General disorders) | 14 | 20
Neutropenic Fever (Blood and lymphatic system disorders) | 14 | 9
Infection (Infections and infestations) | 17 | 18
Nausea / Emisis (Gastrointestinal disorders) | 7 | 13
Neuropathy (Nervous system disorders) | 21 | 14
Rash / Pruitius (Skin and subcutaneous tissue disorders) | 10 | 18
Neutropenia (Blood and lymphatic system disorders) | 67 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 14
Anemia (Blood and lymphatic system disorders) | 10 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2001-05-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT00577993/Prot_SAP_ICF_000.pdf